CLINICAL TRIAL: NCT00278668
Title: Serotonin Uptake to Lymphocytes and Citalopram Platelets Binding of Treatment-Resistant Schizophrenia Patients Before and After Electroconvulsive Therapy
Brief Title: ECT Schizophrenia Serotonin Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Other Study IDs: 123.ctil
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
We suggest to investigate serotonin uptake in schizophrenia patients receiving ECT

DETAILED DESCRIPTION:
We suggest to investigate serotonin uptake in schizophrenia patients receiving ECT

ELIGIBILITY:
Inclusion Criteria:

Participants must meet DSM-IV criteria for schizophrenia, as assessed by the Structured Clinical Interview - Patient Version (SCID) (First et al., 1995).

Ages 18 -55 Men and/or women -

Exclusion Criteria:

1. History of neurological disorders, active substance abuse in the previous 3 months.
2. Estimated IQ less then 70.
3. SSRIs treatment 4 weeks prior to the study.
4. Any subject suffering from inflammatory fever disease will be excluded from the study.

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-10; Study Completion 2006-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Avi Peled, MD, Principal Investigator — Shaar Menashe MHC; Ilan Modai, M.D. MHA, Principal Investigator — Shaar Menashe; Moshe Rehavi, Ph.D., Principal Investigator — TAU